CLINICAL TRIAL: NCT02900729
Title: A Prospective Multicenter Randomized Controlled Trial of Efficacy and Safety of Renal Denervation for Resistant Hypertension
Brief Title: Randomized Controlled Trial of Renal Denervation for Resistant Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai WiseGain Medical Devices Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WiseGo-CT-1601
Record Dates: First submitted 2016-09-07; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Catheter Ablation; Amlodipine; Losartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Denervation plus Medications (Experimental): Renal denervation procedure after randomization plus maintenance of baseline standardised triple anti-hypertensive medications for 90 days and then medically necessary adjustment of antihypertensive medications for another 90 days
  Interventions: Device: Radiofrequency ablation catheter; Drug: Amlodipine, losartan potassium and hydrochlorothiazide
- Medications (Active Comparator): Maintenance of baseline standardised triple antihypertensive medications after randomization for 90 days and then medically necessary adjustment of antihypertensive medications for another 90 days, after which, subjects will be allowed to cross over to perform renal denervation if they still meet the inclusion criteria for the study.
  Interventions: Drug: Amlodipine, losartan potassium and hydrochlorothiazide

INTERVENTIONS:
Device: Radiofrequency ablation catheter — Subjects will be treated with the renal denervation procedure using WiseGo Catheter System after randomization.
  Arms: Renal Denervation plus Medications
Drug: Amlodipine, losartan potassium and hydrochlorothiazide — Standardised triple anti-hypertensive medications of amlodipine 5 mg per day, losartan potassium 50 mg and hydrochlorothiazide 12.5 mg per day in the first 90 days after randomization. Subjects will be allowed to adjust baseline antihypertensive medications where clinically necessary in the second 90 days after randomization.

SUMMARY:
Hypertension represents a significant global public health problem, contributing to vascular and renal morbidity, cardiovascular mortality, and economic burden. For a mostly asymptomatic disease, there is a huge challenge to maintain a good adherence and longtime persistence of drug use so as to adequately control it. Even so, a significant proportion of patients will develop resistant hypertension. In recent years, renal denervation has been argued as an effective means to address blood pressure problem in several non-Chinese clinical trials. The technique is to deliver low level radiofrequency energy through the renal artery wall to target the sympathetic nervous system and then modulate blood pressure.

Shanghai WiseGain Medical Devices Co., LTD has developed the WiseGo Catheter System, which is an irrigated radiofrequency ablation Catheter. With this Catheter, it is expected to improve blood pressure status among patients with resistant hypertension failing polypharmacy. The purpose of this randomized control trial is to obtain an assessment of the efficacy and safety of WiseGo renal denervation technique in the presence of three standard antihypertensive medications in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with primary hypertension has 24-hour ambulatory systolic blood pressure ≥ 135 mmHg and office systolic blood pressure ≥ 140 mmHg /office diastolic blood pressure ≥ 90 mmHg after a 4-week standardised triple therapy.
2. Subject is ≥ 18 and < 80 years old at time of randomization.
3. Subject agrees to have all study procedures performed, and willing to provide written informed consent to participate in this clinical study.

Exclusion Criteria:

1. Subject has acute or serious systemic infection.
2. Subject has a history of renal artery interventional therapy.
3. Subject lacks suitable renal artery anatomy for percutaneous renal sympathetic nerve radiofrequency ablation surgery, including not limited to a presence of serious aorta or renal-artery tortuosity or renal-artery stenosis.
4. Subject has experienced a myocardial infarction, unstable angina pectoris, syncope, or a cerebrovascular accident within three months of the screening period, or has widespread atherosclerosis, with documented intravascular thrombosis.
5. Subject has aortic dissection aneurysm.
6. Subject has primary pulmonary hypertension.
7. Subject has an estimated glomerular filtration rate of less than 40 mL/min/1.73m² according to Modification of Diet in Renal Disease formula.
8. Subject had a definite diagnose of coronary heart disease requiring beta blockers
9. Subject has a Class III - IV of heart failure or left ventricular ejection fraction <45%.
10. Subject had atrial fibrillation.
11. Subject has a significant bleeding tendency or blood system disease(s).
12. Subject has a malignancy or end-stage disease(s).
13. Subject has secondary hypertension.
14. Subject has type 1 diabetes mellitus.
15. Subject has other conditions inappropriate for participation at the investigator's discretion.
16. Subject has a medical ethics of concern at the investigator's discretion, such as a presence of 24-hour Ambulatory Blood Pressure Monitoring average systolic blood pressure ≥ 170 mmHg after a 4-week standardised triple therapy.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-08 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change in average 24-hour systolic blood pressure by ambulatory blood pressure monitoring from baseline | 3 months post-randomization

SECONDARY OUTCOMES:
Incidence of achieving target blood pressure | 6 months post-randomization
  Target blood pressure is defined as daytime ambulatory blood pressure <135/85mmHg, nighttime ambulatory blood pressure <120/70mmHg or average 24-hour ambulatory blood pressure <130/80mmHg, respectively
Change in daytime and nighttime ambulatory systolic blood pressure from baseline | 3 months post-randomization
Change in 24 hour average, daytime and nighttime ambulatory diastolic blood pressure from baseline | 3 months post-randomization
Change in serum creatinine from baseline | 6 months post-randomization
Incidence of adverse event | Through study completion, up to 6 months

OTHER OUTCOMES:
Change in 24 hour average, daytime and nighttime ambulatory systolic/diastolic blood pressure from baseline | 6 months post-randomization
Change in office systolic/diastolic blood pressure from baseline | 6 months post-randomization
Change in patient-recorded home systolic/diastolic blood pressure from baseline | 6 months post-randomization
Incidences of achieving reductions of ≥ 5 mmHg, ≥ 10 mmHg, ≥15 mmHg, and ≥ 20 mmHg in blood pressure, including ambulatory, office and home blood pressure | 6 months post-randomization
Incidences of substantially adjusting antihypertensive medications | 6 months post-randomization
  A substantial adjustment of antihypertensive medications is defined as any changes in number of antihypertensive medications, or type of antihypertensive medications, or ≥ 50% dose change in any ongoing antihypertensive medications in the last two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Dr., Principal Investigator — Zhongshan Hospital affiliated to Fu Dan University
Locations (13):
- China (13):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongshan Hospital affiliated to Fu Dan University, Shanghai, Shanghai Municipality
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Putuo Hospital affiliated to Shanghai Traditional Chinese Medicine University, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Tongji Hospital affiliated to Tongji University, Shanghai, Shanghai Municipality
  - Xinhua Hospital affiliated to Shanghai Jiao Tong University School of Medicine Chongming Branch, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital affiliated to Zhejiang University, Hangzhou, Zhejiang
  - The Second Hospital affiliated to Zhejiang University, Hangzhou, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang
  - The First Hospital affiliated to Wenzhou Medical College, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939
- [Derived] Liu Z, Shen L, Huang W, Zhao X, Fang W, Wang C, Yin Z, Wang J, Fu G, Liu X, Jiang J, Zhang Z, Li J, Lu Y, Ge J. Efficacy and safety of renal denervation for Chinese patients with resistant hypertension using a microirrigated catheter: study design and protocol for a prospective multicentre randomised controlled trial. BMJ Open. 2017 Sep 1;7(9):e015672. doi: 10.1136/bmjopen-2016-015672. PMID 28864691